CLINICAL TRIAL: NCT02224547
Title: Phase II Protocol for Risk-adapted Stereotactic Body Radio Therapy for Stage T1-T3N0 Non-Small Cell Lung Carcinoma
Brief Title: Risk-adapted Stereotactic Body Radiotherapy for Early Non-Small Cell Lung Cancer Using the VERO Stereotactic Body Radio Therapy System
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Christine Collen, MD., Radiaton Oncologist, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lung Vero SBRT
Record Dates: First submitted 2014-05-27; First posted 2014-08-25 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Non-Small Cell Lung Carcinoma
Keywords: non-small cell lung cancer; lung carcinoma; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiotherapy (Experimental): For centrally located T1 and T2 lesions 4 x 12 Gy over 2 weeks will be delivered. Lesions located peripherally will be treated with 3 x 17 Gy, also delivered within 2 weeks. For both schedules, there should be a minimum of 40 hours and a maximum of 8 days between 2 separate fractions. There should be a maximum of 2 fractions per week.
  Interventions: Radiation: Radiotherapy (Fractionated stereotactic body radiation)

INTERVENTIONS:
Radiation: Radiotherapy (Fractionated stereotactic body radiation) — Radiation: Fractionated stereotactic body radiation therapy For centrally located T1 and T2 lesions 4 x 12 Gy over 2 weeks will be delivered. Lesions located peripherally will be treated with 3 x 17Gy, also delivered within 2 weeks. For both schedules, there should be a minimum of 40 hours and a maximum of 8 days between 2 separate fractions. There should be a maximum of 2 fractions per week.

SUMMARY:
The purpose of this study is to perform prospective data analysis on tumor response in terms of local tumor control after 2 years, potential acute and late toxicity and survival in patients with non-metastatic, non-small-cell lung cancer treated by radiotherapy that are medically inoperable due to coexisting comorbidities or that refuse surgery. SBRT regimens used will be 4 fractions of 12 Gy or 3 fractions of 17 Gy depending on tumor location in a risk-adapted approach.

ELIGIBILITY:
Inclusion Criteria:

1. Stage T1,T2,T3N0M0 NSCLC, histological confirmation either by biopsy or cytology
2. Maximal tumor diameter of 6 cm
3. Only T3 lesions based upon thoracic wall involvement, only 1 lesion
4. Informed consent is required
5. Life expectancy of at least 6 months
6. Age >/= 18 y.
7. Karnofsky score ≥ 70 or ECOG score ≤ 2
8. Inoperable patients or patients refusing surgery
9. Patients with measurable lesion (according to RECIST criteria)

Exclusion Criteria:

1. Diagnosis of small cell lung cancer
2. Lymph node involvement
3. Prior radiotherapy to the chest and/or mediastinum
4. No chemotherapy and/or targeted treatment within 3 months before SBRT
5. Pregnant or lactating women
6. Known allergy for CT contrast
7. No FDG-PET
8. Mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study.
9. Patient unlikely to comply with protocol, i.e., uncooperative attitude, inability to return for follow-up visits, extreme degradation of lung function tests and patients not likely to complete the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Toxicity of grade 3+ as assessed by NCI CTCAE v4.0 | From start of SBRT until 1 year. After 1 year until end of follow-up for late toxicity
  To monitor potential toxicity in patients with stage T1,T2,T3 N0 non-small cell lung carcinoma (NSCLC), treated with primary stereotactic body radiation therapy (SBRT)

SECONDARY OUTCOMES:
Time to local progression | every 3 months for the first 2 years. From 3 to 5 years every 6 months. After From start of SBRT until date of death, regional fialure of last follow-up. Aanalysis occurs when all patients have been potentially followed for 24 months.
  Overall survival, local progression free survival, disease free survival, time from start of SBRT to death, local, regional or disseminated recurrence.

OTHER OUTCOMES:
Quality of life | baseline at inclusion, at 1 month-, 3 months- and 12 months from start SBRT
  Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Christine Collen, MD, Principal Investigator — UZ Brussel Radiotherapie dienst
Locations (1):
- UZ Brussel Radiotherapie dienst, Jette, Brussels Capital, Belgium

REFERENCES:
- [Derived] Levy A, Guckenberger M, Hurkmans C, Nestle U, Belderbos J, De Ruysscher D, Faivre-Finn C, Le Pechoux C. SBRT Dose and Survival in Non-Small Cell Lung Cancer: In Regard to Koshy et al. Int J Radiat Oncol Biol Phys. 2015 Jul 15;92(4):945-6. doi: 10.1016/j.ijrobp.2015.03.032. No abstract available. PMID 26104945